CLINICAL TRIAL: NCT02738398
Title: Optimizing Lung Cancer Nodal Staging With FDG PET/CT Through Improved Image Acquisition and Reconstruction
Brief Title: FDG PET/CT in Lung Cancer Staging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UPCC 20515
Record Dates: First submitted 2016-04-12; First posted 2016-04-14 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET imaging (Experimental): PET imaging
  Interventions: Radiation: FDG PET/CT

INTERVENTIONS:
Radiation: FDG PET/CT

SUMMARY:
Prospective study of the effects of image acquisition and reconstruction parameters on accuracy of FDG PET/CT mediastinal nodal staging in NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, at least 18 years of age
* Patients with NSCLC diagnosis who have been referred for a clinical FDG PET/CT staging scan as part of their standard of care
* Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Inability to tolerate additional imaging time in the opinion of the investigator or treating physician.
* Only individuals (aged 18 or over) who can understand and give informed consent will be eligible to participate in this study. Individuals who are considered to be mentally disabled will not be recruited for this study. All subjects must be able to give informed consent. We will not be using specific methods to assess decisional capacity. Economically disadvantaged persons will not be vulnerable to undue influence, as this study offers no compensation and there is no additional cost associated with the additional study imaging time. All individuals will be told that their choice regarding study participation will in no way change their access to clinical care or their ability to undergo the standard clinical FDG PET/CT scan. This should negate any undue influence or coercion. Children, fetuses, neonates, or prisoners are not included in this research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pryma, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States